CLINICAL TRIAL: NCT01206413
Title: A Randomized Clinical Trial of Home-based Exercise Combined With a Slight Caloric Restriction on Obesity Prevention Among Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Mauro Felippe Felix Mediano, State University of Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNPQ500404/2003-8
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Obesity Prevention
Keywords: overweight; treatment; women
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LGI (Experimental): Low glycemic index
  Interventions: Dietary Supplement: Low glycemic index diet
- HGI (Active Comparator): High glycemic index
  Interventions: Dietary Supplement: High glycemic index diet
- HB (Experimental): Home-based exercise
  Interventions: Other: Home-based exercise intervention
- CONTROL (Active Comparator): Non-exercisers
  Interventions: Other: Non-exercisers

INTERVENTIONS:
Dietary Supplement: Low glycemic index diet
  Arms: LGI
Dietary Supplement: High glycemic index diet
  Arms: HGI
Other: Home-based exercise intervention
  Arms: HB
Other: Non-exercisers
  Arms: CONTROL

SUMMARY:
The study investigated the effectiveness of home-based exercise combined with a slight caloric restriction on weight change during 12 months in non-obese women. In addition the investigators evaluate the effects of baseline insulin resistance on modulation of weight change.

A randomized clinical trial with a factorial design was conducted from 2003 to 2005. Two hundred three middle-aged women (Rio de Janeiro/Brazil), 25-45 years, were randomly assigned to one of two groups: control (CG) and home-based exercise (HB). The HB group received a booklet on aerobic exercise that could be practiced at home (3 times/week - 40 min/session), in low-moderate intensity, during 12 months. Both groups received dietary counseling aimed at a slight energy restriction of 100-300 calories per day.

The HB experienced a greater weight loss in the first 6 months (-1.4 vs. -0.8 kg; p=0.04), but after 12 months there was no differences between groups (-1.1 vs. -1.0; p=0.20). Of the serum biochemical markers, HDL-cholesterol showed major change, with an increase at month 12 of 18.3 mg/dl in the HB compared to 9.5 in the CG (p<0.01). At baseline the non-IR group (n=121) compared to IR (n=64) had similar values of BMI (26.7 vs. 26.3 p=0.21), but statistically significant lower values of waist, glucose, insulin and HOMA-IR, as expected. When the group non-IR and IR were further stratified by GI diet, there were no differences according to diet in both groups. Women classified as IR at baseline had greater weight loss after 12 months of follow-up (-1.62 kg vs. -1.08 kg; p=0.01), and HB exercise helped to reduce weight only among NIR women (-1.51 vs. -0.68; p=0.04); no differences were observed between intervention groups for IR women (-1.54 vs. -1.66; p=0.24). There were no differences between IR and NIR groups for lipid profile after adjustment for weight changes. During follow-up, changes were more pronounced among those women in the high GI diet. These differences were statistically significant for weight and BMI and were greater among the IR compared to the non-IR. Changes in HOMA-IR after 3 months of follow-up were different comparing non-IR with IR at baseline. The IR had a reduction in the HOMA-IR, whereas in the non-IR this value increased (-0.73 vs. +0.37; p=<0.001). Also this reduction was greater among high compared to low GI diet (p=0.04).

ELIGIBILITY:
Inclusion Criteria:

Non-obese women aged 25-45 years

Exclusion Criteria:

Physician-diagnosed thyroid disease or diabetes or who were menopausal or any other disease that could be influenced by intervention

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2003-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

REFERENCES:
- [Derived] Mediano MF, Neves FA, Cunha AC, Souza EP, Moura AS, Sichieri R. Changes in body weight, C-reactive protein, and total adiponectin in non-obese women after 12 months of a small-volume, home-based exercise program. Clinics (Sao Paulo). 2013;68(8):1121-7. doi: 10.6061/clinics/2013(08)10. PMID 24037008